CLINICAL TRIAL: NCT05028348
Title: A Phase 3 Randomized, Open-label Trial of Selinexor, Pomalidomide, and Dexamethasone (SPd) Versus Elotuzumab, Pomalidomide, and Dexamethasone (EloPd) in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of Combination of Selinexor, Pomalidomide, and Dexamethasone (SPd) Versus Elotuzumab, Pomalidomide, and Dexamethasone (EloPd) in Subject With Previously Treated Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN29
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; elotuzumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selinexor, pomalidomide and dexamethasone (SPd) (Experimental): Selinexor will be given as an oral dose:
  40 mg (2 20 mg tablets) once weekly (QW) on Days 1, 8, 15, and 22 of each 28-day cycle.
  * Pomalidomide will be given as an oral 4 mg dose QD on Days 1 to 21 of each 28-day cycle.
  * Patients ≤75 years:
    o Dexamethasone will be given as an oral 40 mg dose QW on Days 1, 8, 15, and 22 of each 28-day cycle. Dose may be divided over 2 days at the Investigator's discretion.
  * Patients > 75 years:
    * Dexamethasone will be given as an oral 20 mg dose QW on Days 1, 8, 15, and 22 of each 28-day cycle. Dose may be divided over 2 days at the Investigator's discretion.
  Interventions: Drug: Selinexor; Drug: Pomalidomide; Drug: Dexamethasone Oral
- Elotuzumab, Pomalidomide and Dexamethasone (EloPd) (Active Comparator): Elotuzumab will be given IV 10 mg/kg on Days 1, 8, 15, and 22 of cycle 1 and 2 then 20 mg/kg on Day 1 of cycles ≥3 of each 28-day cycle.
  * Pomalidomide will be given as an oral 4 mg dose once a day (QD) on Days 1 to 21 of each 28-day cycle.
  * Patients ≤75 years:
    * Dexamethasone 28 mg PO + 8 mg IV on days of elotuzumab dosing
    * Dexamethasone 40 mg PO on non-elotuzumab days (e.g., days 8, 15, and 22 of cycle 3 and beyond). Dose may be divided over 2 days at the Investigator's discretion.
  * Patients >75 years:
    * Dexamethasone 8 mg PO + 8 mg IV on days of elotuzumab dosing
    * Dexamethasone 20 mg PO on non-elotuzumab dosing weeks (e.g., days 8, 15, and 22 of cycle 3 and beyond). Dose may be divided over 2 days at the Investigator's discretion.
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Selinexor — Selinexor will be given as an oral dose 40 mg (2 20 mg tablets) QW on Days 1, 8, 15, and 22 of each 28-day cycle.
  Other Names: KPT-330
  Arms: Selinexor, pomalidomide and dexamethasone (SPd)
Drug: Elotuzumab — Elotuzumab will be given IV 10 mg/kg on Days 1, 8, 15, and 22 of cycle 1 and 2 then 20 mg/kg on Day 1 of cycles ≥3 of each 28-day cycle.
  Arms: Elotuzumab, Pomalidomide and Dexamethasone (EloPd)
Drug: Pomalidomide — Pomalidomide will be given as an oral 4 mg dose QD on Days 1 to 21 of each 28-day cycle.
Drug: Dexamethasone Oral — Dexamethasone will be given as an oral 40 mg dose QW on Days 1, 8, 15, and 22 of each 28-day cycle. Preferred dosing of dexamethasone is 40 mg QW for patients who are ≤75 years of age (20 mg QW for >75-year-old patients at the Investigator's discretion) before QW dosing of selinexor, however, it may be divided over 2 days at the Investigator's discretion.

SUMMARY:
This phase 3 randomized, open-label multicenter trial will compare the efficacy, safety and the impact on health-related quality of life (HR-QoL) of SPd versus EloPd in pomalidomide-naïve patients with MM who have received 1 to 4 prior anti-MM regimens and been treated with an immunomodulatory imide drug (IMiD), proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody (mAb).

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory MM with measurable disease per IMWG guidelines as defined by at least 1 of the following:

   1. Serum M-protein ≥0.5 g/dL (≥5 g/L) by serum protein electrophoresis (SPEP) or, for immunoglobulin (Ig) A or D myeloma, by quantitative serum IgA or IgD levels ≥ 0.5 g/dL.
   2. Urinary M-protein excretion ≥200 mg/24 hours
   3. Serum free light chain (FLC) ≥100 mg/L, provided that the FLC ratio is abnormal (normal FLC ratio: 0.26 to 1.65)
2. Received at least 1 and no more than 4 prior anti-MM lines of therapy. Induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 line of therapy.
3. Prior therapy that includes ≥ consecutive cycles of lenalidomide and a proteasome inhibitor given alone or in combination
4. Prior therapy with an anti-CD38 mAb as part of their immedicate last treatment prior to study entry (Before protocol version2.0, patient with any prior therapy with an anti-CD38 mAb were eligible for the study).
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
6. Resolution of any clinically significant non-hematological toxicities (if any) from previous treatments to Grade ≤1 by Cycle 1 Day 1 (C1D1). Patients with Grade 2 non-hematological toxicities may be included.
7. Adequate hepatic function within 28 days prior to C1D1:

   1. Total bilirubin <2 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of <3 × ULN)
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 × ULN
8. Adequate renal function within 28 days prior to C1D1 (estimated creatinine clearance [CrCl] of ≥15 mL/min (not requiring dialysis), calculated using the formula of Cockcroft and Gault or measured by 24-hour urine collection).
9. Adequate hematopoietic function within 7 days prior to C1D1 defined as absolute neutrophil count ≥1.5 x 109/L , hemoglobin ≥8.5 g/dL, and platelet count ≥100 x 109/L (patients for whom <50% of bone marrow nucleated cells are plasma cells) or ≥75 x 109/L (patients for whom ≥50% of bone marrow nucleated cells are plasma cells).

   1. Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (e.g., eltrombopag, romiplostim, or interleukin-11) must have a 2-week interval between growth factor support and the Screening assessments, but they may receive growth factor support during the study.
   2. Patients must have:

      * At least a 2-week interval from the last red blood cell (RBC) transfusion prior to the Screening hemoglobin assessment, and
      * At least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment.

   However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
10. Patients with active hepatitis B virus (HBV) are eligible if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/mL. Patients with evidence of non-active HBV should be discussed with the Medical Monitor and should be monitored or receive prophylaxis at the discretion of the Investigator and study site institutional guidelines
11. Patients with a history of hepatitis C virus (HCV) are eligible if they have received adequate curative anti-HCV treatment and HCV viral load is below the limit of quantification.
12. Patients with a history of human immunodeficiency virus (HIV) are eligible if they have CD4+ T cell counts ≥350 cells/µL, negative viral load, and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year and should be on established antiretroviral therapy (ART) for at least 4 weeks.
13. Female patients of childbearing potential must have a negative serum pregnancy test within 10 to 14 days and a second test within 24 hours prior to the first dose of study treatment. Female patients of childbearing potential and fertile male patients who are sexually active must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.
14. Age ≥18 years at the time of signing informed consent.
15. Written informed consent signed in accordance with federal, local, and institutional guidelines.
16. Patients must be able and willing to take enteric-coated aspirin according to clinical practice, or if history of prior thrombotic disease, must be fully anticoagulated with warfarin (international normalized ratio [INR] 2-3) or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism (PE) at the Investigator's discretion. For patient on warfarin, INR should be repeated as clinically indicated. Use of alternative anticoagulants, such as direct oral anticoagulants, may be considered per Investigator discretion.

Exclusion Criteria:

1. Smoldering MM.
2. Plasma cell leukemia.
3. Documented active systemic amyloid light chain amyloidosis.
4. Any history of central nervous system MM.
5. Prior treatment with:

   1. A selective inhibitor of nuclear export (SINE) compound, including selinexor
   2. Pomalidomide and/or elotuzumab.
6. Any concurrent medical condition or disease that is likely to interfere with study procedures.
7. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to C1D1. Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
8. Known intolerance, hypersensitivity, or contraindication to any of the study treatments.
9. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy including investigational therapies and high dose dexamethasone (i.e., 40 mg daily for 4 days per week) ≤2 weeks prior to C1D1. Patients on long-term glucocorticoids during Screening do not require a washout period but must be able to tolerate the specified dexamethasone dose in this study.
10. Prior autologous stem cell transplantation <60 days or allogeneic stem cell transplantation <4 months prior to C1D1.
11. Major surgery within 4 weeks prior to C1D1.
12. Active graft versus host disease after allogeneic stem cell transplantation.
13. Pregnant or breastfeeding females.
14. In the opinion of the Investigator, patients who are below their ideal body weight and would be unduly impacted by changes in their weight.
15. Clinically significant cardiac disease, including:

    1. Myocardial infarction within 6 months before C1D1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
    2. Uncontrolled cardiac arrhythmia (CTCAE v. 5.0 Grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
    3. Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
16. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
17. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
18. Contraindication to any of the required concomitant drugs or supportive treatments.
19. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | from randomization to the date of disease progression or death (approximately up to 5 years)
  from date of randomization until the date of first confirmed progressive disease (PD), per IMWG response criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | from screening until end of treatment/progressive disease (approximately up to 2 years)
  defined as any response ≥PR (i.e., PR [partial response], VGPR [very good partial response], CR ([complete response], or sCR [stringent complete response])
Overall survival (OS) | From randomization until death from any cause (up to 3 years after end of treatment)
  Overall Survival
Duration of response | screening, Day 1 of each treatment cycle (each cycle is 28 days), at end of treatment, and every 3 months up to 3 years
  Duration of response (PR or better), duration of CR, duration of sCR, and duration of minimal residual disease (MRD) -negative status, are calculated from the date of the initial documentation of a response (PR or better), or CR or better, or sCR, or MRD-negative status to the date of the first documented evidence of disease progression, as defined in the IMWG criteria, whichever occurs first.
Time to response | screening, Day 1 of each treatment cycle (each cycle is 28 days), at end of treatment, and every 3 months up to 3 years
  Time to response (PR or better), time to CR/sCR are defined as the time from randomization to date of initial response (or initial CR/sCR)
Progression-free survival on the next line of therapy (PFS2) | the time from randomization to progression on the next line of treatment or death, whichever comes first., assessed up to approx. 5 years
  Progression-free survival on the next line of therapy (PFS2) is defined as the time from randomization to progression on the next line of treatment or death, whichever comes first.
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core module (EORTC QLQ-C30) score and the difference between-treatment arms | screening, Day 1 of each treatment cycle (each cycle is 28 days), at end of treatment (up to 2 years)
  The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-of-Life (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.
Change in EORTC QLQ- 20-item Multiple Myeloma module (MY-20) score and the difference between-treatment arms | screening, Day 1 of each treatment cycle (each cycle is 28 days), at end of treatment (approximately up to 2 years)
  The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in subjects with MY. The module comprises 20 questions that address four myeloma-specific HRQoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspective, and Body Image. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.
EQ-5D-5L health utility values and the difference between-treatment arms | screening, Day 1 of each treatment cycle (each cycle is 28 days), at end of treatment (approximately up to 2 years)
  The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today"
safety and tolerability of SPd versus EloPd in patients with RRMM | continuously from screening untill 30 days after last study treatment. (approximately up to 2 years)
  Safety and tolerability of study treatment will be evaluated based on occurrence, nature and severity of adverse events as categorized by the Common Terminology Criteria of Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (20):
- France (3):
  - CHRU Hôtel Dieu, Nantes
  - CHU Hôpital Saint Antoine, Paris
  - La Pitié, Paris
- Germany (4):
  - Klinikum Chemnitz, Chemnitz
  - Marien Hospital Dusseldorf, Düsseldorf
  - University Medicine Greifswald, Medical Clinic and Polyclinic for Internal Medicine, Greifswald
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
- Alexandra General Hospital -Department of Clinical Therapeutics N.K. Univ. of Athens, Athens, Greece
- Spain (12):
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala D Oncolocia Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital de Cabueñes, Gijón
  - Institut Català D'Oncologia - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario 12 de Octubre, Madrid
  - H. General Universitario Morales Meseguer, Murcia
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - H. Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - H.U. La Fe, Valencia